CLINICAL TRIAL: NCT05750537
Title: Enhanced Multicomponent Proactive Navigator-Assisted Cessation of Tobacco Use in Low-Income Patients
Acronym: EMPACT-Us
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Family Health Centers of San Diego (Other)
Collaborators: University of California, San Diego (Other); Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T32CF4745
Record Dates: First submitted 2023-02-07; First posted 2023-03-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Use Cessation
Keywords: Tobacco Use Cessation; FQHC; San Diego; Electronic Health Record; EHR; Kick It California; FHCSD; UCSD; Family Health Centers of San Diego; University of California San Diego; California; Southern California; Low-income populations; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMPACT-Us (Experimental): An innovative suite of tobacco cessation services designed in partnership with patients, providers, and other community stakeholders during a pilot study.
  Interventions: Behavioral: EMPACT-Us
- Newly-enhanced usual care (EUC) (No Intervention): Newly-enhanced usual care (EUC)

INTERVENTIONS:
Behavioral: EMPACT-Us — A suite of tobacco cessation services supported by patient navigation designed in close partnership with patients, providers, and community stakeholders.
  Arms: EMPACT-Us

SUMMARY:
This research study is being conducted to test the effectiveness of the Enhanced Multicomponent Proactive Navigator-Assisted Cessation of Tobacco Use (EMPACT-Us), an innovative suite of tobacco cessation services designed in partnership with patients, providers, and other community stakeholders during a pilot study.

We hypothesize that EMPACT-Us will be more effective than the newly-enhanced usual care on improving engagement in tobacco treatments, quit attempts and biochemically verified cessation at 6-and 12-months post initial offerings.

DETAILED DESCRIPTION:
The investigators propose a stepped-wedge cluster randomized trial. Eight of the largest FHCSD clinics with geographic distribution covering a wide region of San Diego were selected. Based on chart review, the investigators estimate that there are 13,496 tobacco users who are active patients at the selected clinics and could present to one or more clinics during the study period. This population represents roughly 70% of the tobacco users at FHCSD. The larger clinics are chosen based on size, special populations represented, and staff size. The study duration was divided into five 6-month periods. After a baseline period, four pairs of clinics (8 total clinics) will be assigned randomly to begin the active treatment at one of the four subsequent periods. No other clinic characteristics are used for randomization. Tobacco users first tobacco-related visit will anchor subsequent assessments of tobacco use and engagement in tobacco treatments within their electronic medical records and in surveys during the duration of the study.

Activities are designed to evaluate tobacco treatments within FHCSD and to generalize these evaluations to other health clinics serving similar low-income communities. Activities are organized within the Milestones, each building upon the other, leading to the ultimate test of two workflows offering a suite of tobacco cessation services. Milestone 1 (1-6mo) includes startup and training (TE Coach curriculum adaptation, MA training, Primary Care Provider (PCP) training) and baseline data collection using system-level infrastructure assessment and rapid, iterative improvement; Milestone 2 (6-33mo) includes the testing of EMPACT-Us suite of services, with evaluation and fidelity checks built into implementation through Milestone 3 (4-33mo.), which will include conducting qualitative semi-structured interviews and surveys designed to understand the experiences of patients, N-MAs, PCPs, and TE Coaches. Staff will be interviewed either in person or remotely, while patients will be offered surveys either remotely over the phone or via email or SMS beginning two to four weeks after their index visit.; Milestone 4 (7-35mo) data analysis weaves through most of the study to inform work as the investigation progresses; and Milestone 5 (6-36mo) manuscript preparation and dissemination, is planned throughout the study period and beyond.

For the current project, UC San Diego investigators and staff are engaged with FHCSD in delivering the intervention that the investigators partnered to develop. While primarily housed at UC San Diego, this project will include regular onsite interactions with clinical records, individual interviews, interacting with FHCSD providers and viewing clinical information in both clinical intervention training and evaluation roles that again will include contact with patient PHI. The investigators will be removing PHI prior to final qualitative and quantitative analyses and reporting results using de-identified data.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco user
* 18 years old
* Speaks English or Spanish

No exclusions due to:

* Nationality
* Mental health status
* Substance use
* Race
* Sexual orientation
* Ethnicity

Inclusion into saliva collection:

* Met level 1 criteria for inclusion into study
* Reports abstinence at follow-up assessment

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a lung cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13496 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Engagement with tobacco-use treatment as captured through Electronic Health Record queries | 7 to 35 months
  Engagement with tobacco use treatment is defined as at least one dose/session of evidence-based pharmacotherapy or behavioral counseling for smoking cessation using the EHR.
Tobacco-use quit attempts as assessed through Electronic Health Record queries | 7 to 35 months
  Quit attempts are defined as the stated intention to achieve long-term cessation and an ability to refrain smoking evidenced by a self-reported 24-hour period of no smoking. ((e.g. C-TUQ: How long has it been since you last smoked a cigarette (even one or two puffs)?))
Biochemically verified tobacco-use cessation as assessed through cotinine saliva test | 6 and 12 months
  Tobacco-use cessation is defined as prolonged abstinence at the 6- and 12- month follow periods, biochemically verified through cotinine saliva tests.

CONTACTS AND LOCATIONS:
Overall Officials: David Strong, BA, MS, PhD, Principal Investigator — University of California, San Diego; Karim Ghobrial-Sedky, MD, MSc, DFAPA, Principal Investigator — Family Health Centers of San Diego
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Family Health Centers of San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flocke SA, Vanderpool R, Birkby G, Gullett H, Seaman EL, Land S, Zeliadt S. Addressing Tobacco Cessation at Federally Qualified Health Centers: Current Practices & Resources. J Health Care Poor Underserved. 2019;30(3):1024-1036. doi: 10.1353/hpu.2019.0071. PMID 31422986
- [Background] Flocke SA, Seeholzer E, Lewis SA, Gill IJ, Rose JC, Albert E, Love TE, Kaelber D. 12-Month Evaluation of an EHR-Supported Staff Role Change for Provision of Tobacco Cessation Care in 8 Primary Care Safety-Net Clinics. J Gen Intern Med. 2020 Nov;35(11):3234-3242. doi: 10.1007/s11606-020-06030-7. Epub 2020 Jul 23. PMID 32705473
- [Background] Fernandez ME, Schlechter CR, Del Fiol G, Gibson B, Kawamoto K, Siaperas T, Pruhs A, Greene T, Nahum-Shani I, Schulthies S, Nelson M, Bohner C, Kramer H, Borbolla D, Austin S, Weir C, Walker TW, Lam CY, Wetter DW. QuitSMART Utah: an implementation study protocol for a cluster-randomized, multi-level Sequential Multiple Assignment Randomized Trial to increase Reach and Impact of tobacco cessation treatment in Community Health Centers. Implement Sci. 2020 Jan 30;15(1):9. doi: 10.1186/s13012-020-0967-2. PMID 32000812
- [Background] Fiore M, Adsit R, Zehner M, McCarthy D, Lundsten S, Hartlaub P, Mahr T, Gorrilla A, Skora A, Baker T. An electronic health record-based interoperable eReferral system to enhance smoking Quitline treatment in primary care. J Am Med Inform Assoc. 2019 Aug 1;26(8-9):778-786. doi: 10.1093/jamia/ocz044. PMID 31089727
- [Background] Levinson AH, Valverde P, Garrett K, Kimminau M, Burns EK, Albright K, Flynn D. Community-based navigators for tobacco cessation treatment: a proof-of-concept pilot study among low-income smokers. BMC Public Health. 2015 Jul 9;15:627. doi: 10.1186/s12889-015-1962-4. PMID 26155841
- [Derived] Ramirez GF, Badii NZ, Mohn P, Northrup A, Smoot C, Doran N, Brouwer K, Myers M, Godino J, Liu J, Ghobrial-Sedky K, Strong D. Assessing the effects of Enhanced Multicomponent Proactive Navigator-Assisted Cessation of Tobacco Use within a federally qualified health center (EMPACT-Us): a protocol study. BMC Public Health. 2024 Dec 18;24(1):3496. doi: 10.1186/s12889-024-20997-6. PMID 39695566